CLINICAL TRIAL: NCT03941626
Title: EGFRvIII/DR5/NY-ESO-1/Mesothelin CAR-T/TCR-T Cells Immunotherapy for Solid Malignancies
Brief Title: Autologous CAR-T/TCR-T Cell Immunotherapy for Solid Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen BinDeBio Ltd. (Industry)
Collaborators: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019BDB016
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Esophagus Cancer; Hepatoma; Glioma; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Hepatocellular; Glioma; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T/TCR-T cells immunotherapy (Experimental): Enrolled patients will receive CAR-T cell immunotherapy with several different specific Chimeric antigen receptors aiming at different antigens respectively by infusion.
  Interventions: Biological: CAR-T/TCR-T cells immunotherapy

INTERVENTIONS:
Biological: CAR-T/TCR-T cells immunotherapy — According to tumor burden and other conditions, patients will be treated with cyclophosphamide or fludarabine,then,CAR-T cells will be infused 48-72 hours later.

SUMMARY:
This is a single arm, open-label, uni-center, phase I-II study to evaluate the safety and effectiveness of CAR-T/TCR-T cell immunotherapy in treating with different malignancies patients.

DETAILED DESCRIPTION:
The study is a multi-target gene-modified immunotherapy. CAR-T/TCR-T cells include four different tumor-specific antibody.They are as following:anti-NY-ESO-1 antibody foresophagus cancer;anti-DR5 antibody for hepatoma;;anti-EGFR vIII antibody for hepatoma and glioma;anti-Mesothelin antibody for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing to sign an informed consent.
2. Male or female patients aged 18 to 70 years .
3. Estimated survival of ≥ 12 weeks.
4. Pathological sections with positive expression of NY-ESO-1, Mesothelin, EGFRvIII and DR5 was confirmed by biopsy IHC test within 12 months.If NY-ESO-1 is positive expression ,positive HLAA*0201 is required at the same time.
5. Solid tumor must have at least one measureable disease according to RECIST 1.1.
6. Routine blood test#hemoglobin>=90 g/L; platelet>=50×10^9/L.
7. Liver function:ALT and AST≤2.5 times upper limits of normal (If the tumor infiltration is the main cause of abnormal liver function ,ALT and AST≤5 times upper limits of normal); bilirubin<2.0 mg/dL.
8. Renal function:BUN: 9-20mg / dl; serum creatinine≤ 1.5 times upper limits of normal; endogenous creatinine clearance rate≥50 ml/min .
9. Negative serum antibody for EBV, CMV, HIV , syphilis, HBVa nd HCV.
10. Cardiac function: stable hemodynamic and left ventricular ejection fraction (LVEF)>=55%.
11. ECOG score:0-1.
12. Adequate venous access for apheresis, and no other contraindications for leukapheresis .
13. Women of child-bearing age must have evidence of negative pregnancy test. Subjects of reproductive potential must agree to use acceptable birth control methods within 1 year after treatment, as described in protocol.
14. Subjects with hypertension/diabetes must be stable blood pressure/blood glucose or ≤CTCAE 1 level 2 weeks before the screening.

In addition to the above criteria for inclusion, the following criteria shall be met according to the indications:

Patients with glioblastoma：

1. First disease progression or disease recurrence (≥ 1 cm and ≤ 5 cm) of a supratentorial WHO grade IV malignant glioma (GBM or gliosarcoma) based on imaging studies with measurable disease.
2. EGFRvIII, the target antigen, must be identified on tumor tissue by IHC or PCR, i.e. EGFRvIII positive via pathology report.
3. Insensitivity to chemoradiotherapy or chemoradiotherapy failure after operation molecular pathology.
4. Refused to receive radiotherapy or chemotherapy treatment.

Patients with liver cancer

1. DR5 or EGFRvIII positive via pathology report.
2. Untreatable by surgery ; Or postoperative recurrence ;Or no effective treatment.
3. Liver function：child-pugh A grade or child-pugh B grade.

Patients with gastric cancer

1. Mesothelin positive via pathology report.
2. The pathological stage：IIIA～IV.
3. chemoradiotherapy failure
4. Refused or unable to get surgery.

Patients with esophageal cancer

1. NY-ESO-1 positive via pathology report and HLA-A*0201 positive in blood.
2. Refuse or unable to get surgery.
3. Postoperative recurrence or chemoradiotherapy failure.

Exclusion Criteria:

1. ECOG≥2.
2. malignant tumor cells with T cell origin via pathology test.
3. Organ failure: stage III or IV congestive heart failure; Renal failure and uremia; respiratory failure; disturbance of consciousness.
4. Acute or chronic GVHD after allogeneic hematopoiesis; Or being treated for GVHD; Or hormone or immunosuppressant used within 30 days
5. steroid hormoneswere used before and after blood collection and infusion
6. Patients with HIV infection or active hepatitis
7. Uncontrolled active infection.
8. Enrolled to other clinical study in the last 4 weeks.
9. Patients with systemic auto-immune disease or immunodeficiency.
10. Patients with neuropathy or psychosis, including dementia or epilepsy, or history of psychotropic substance abuse, or other substantial lesions that may increase central neurotoxicity.
11. Concomitant with the second tumor or other malignant tumors.
12. Patients with bone metastases are at risk of a pathological fracture resulting in paraplegia or life threatening.
13. Live attenuated vaccine was administered within 4 weeks prior to blood collection.
14. Blood oxygen saturation is maintained by oxygen inhalation.
15. Received major surgery within 2 weeks prior to screening ;Or Plan to receive surgery during study or within 2 weeks after injection.
16. Other patients that researchers considered unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events evaluated with NCI CTC AE, version 4.0 | 48 months
  Safety evaluation

SECONDARY OUTCOMES:
Clinical response | 48 months
  Clinical response to T-cell infusion, especially change of tumor volume will be evaluated by comparing disease identified by computed tomography, magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No